CLINICAL TRIAL: NCT02307357
Title: The Effects of Newcomball Training on Physical Fitness and Mood State of Middle Age Women in Israel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Wingate Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0056-14
Record Dates: First submitted 2014-11-06; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- newcomball players (Experimental): active newcomball women players will perform physical fitness tests
  Interventions: Behavioral: physical fitness tests
- control (Experimental): not physically active women will perform physical fitness tests
  Interventions: Behavioral: physical fitness tests

INTERVENTIONS:
Behavioral: physical fitness tests — the subjects will perform 6 different tests to evaluate their physical fitness

SUMMARY:
Habitual physical activity was found to be positively related to better health and well-being. One of the most popular physical activity forms is ball games. In Israel, there is a growing popularity in a new ball game - Newcomball - which is being played by many middle age, non-athlete, women. However, so far, no study had evaluated the contribution of the game to improvement in the participants' physical fitness. The aim of this study, therefore, is to evaluate the effects of six month two weekly Newcomball training sessions to the physical fitness of middle age women.

DETAILED DESCRIPTION:
Physical fitness will be evaluated by six different physical tests: 1. agility T test, 2. "shuttle run" test for aerobic capacity, 3. vertical jump, 4. power ball throw, 5. "sit and reach" flexibility test , 6. 20 m all-out run speed test.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults women

Exclusion Criteria:

non healthy, using drugs, competitive athletes women-

Ages: 28 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of physical fitness of newcomball players vs. non active women | six month
  we will perform physical fitness tests to 2 groups: newcomball players and non active women in the beginning of games season and in the middle of the season. the measure is:.vertical jump, measured by power plate (in seconds),
Evaluation of physical fitness of newcomball players vs. non active women | six month
  power ball through measures the distance in meters
Evaluation of physical fitness of newcomball players vs. non active women | six month
  agility T-test, measures time to complete the test( in seconds)
Evaluation of physical fitness of newcomball players vs. non active women | six month
  flexibility measures the distance of hands in a sit and reach test (centimeters)
Evaluation of physical fitness of newcomball players vs. non active women | six month
  velocity measures time to complete 20 meters run (seconds)
Evaluation of physical fitness of newcomball players vs. non active women | six month
  aerobic shuttle run test, measures the time and distance completed in graded run test, in which velocity increased until exhaustion (meter and minutes)

CONTACTS AND LOCATIONS:
Overall Officials: sharon tsuk, PhD, Study Director — Wingate Institute
Locations (1):
- Wingate Institute, Netanya, Israel